CLINICAL TRIAL: NCT03028077
Title: The Efficacy and Safety of GS-3K8 and GINst15 on Acute Respiratory Illness in Healthy Subjects
Brief Title: Effects of GS-3K8 and GINst15 on Acute Respiratory Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Soo-Wan Chae, Principal investigator, Clinical Trial Center for Functional Foods, Chonbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CTCF2_2014_GN
Record Dates: First submitted 2017-01-17; First posted 2017-01-23 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Acute Respiratory Infection
Keywords: ultrafiltered red ginseng; hydrolyzed ginseng; acute respiratory illness; clinical trial

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- GS-3K8 (Experimental): GS-3K8 (6 cap/day, 500 mg/cap) for 12 weeks
  Interventions: Dietary Supplement: GS-3K8
- GINst15 (Experimental): GINst15 (6 cap/day, 500 mg/cap) for 12 weeks
  Interventions: Dietary Supplement: GINst15
- Placebo (Placebo Comparator): Placebo for 12 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: GS-3K8 — GS-3K8 (ultrafiltered red ginseng extract) 1 g/day
  Arms: GS-3K8
Dietary Supplement: GINst15 — GINst15 (hydrolyzed ginseng extract) 1 g/day
  Arms: GINst15
Dietary Supplement: Placebo — Placebo 1 g/day
  Arms: Placebo

SUMMARY:
This study was conducted to investigate the effects of daily supplementation of GS-3K8 or GINst15 on acute respiratory illness (ARI) in healthy subjects.

DETAILED DESCRIPTION:
This study was a 8 weeks, randomized, double-blind, placebo-controlled trial. Forty five subjects were randomly divided into GS-3K8 (Ultrafiltered red ginseng extract) or GINst15 (Hydrolyzed ginseng extract) or placebo group. The primary clinical outcome measure was the incidence of ARI. The secondary clinical outcome measure was the development and duration of ARI symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Age 39-65 years with healthy adults

Exclusion Criteria:

* Subjects had been vaccinated against influenza in the previous 6 months
* Subjects with symptoms of upper respiratory tract infection
* Subjects with acute/chronic disease
* History of alcohol or substance abuse
* History of disease that could interfere with the test products or impede their absorption
* Subjects taking medications such as immune or upper respiratory tract infection related drug or functional foods
* Abnormal liver or kidney function tests
* Pregnant or lactating women and heavy smokers
* Being judged by the responsible physician of the local study center as unfit to participate in the study

Ages: 39 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Incidence rate of ARI (by questionnaire) | 18 weeks (intervention for 12 weeks, follow up for 6 weeks after termination)
  Incidence of ARI were assessed before and after intervention and followed up for 6 weeks after termination.

SECONDARY OUTCOMES:
Development of ARI symptoms (by questionnaire) | 18 weeks (intervention for 12 weeks, follow up for 6 weeks after termination)
  Development of ARI symptoms (score) were assessed before and after intervention and followed up for 6 weeks after termination.
Duration of ARI symptoms (by questionnaire) | 18 weeks (intervention for 12 weeks, follow up for 6 weeks after termination)
  Duration of ARI symptoms were assessed before and after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Hwan Hwang, M.D. Ph. D, Principal Investigator — Chonbuk National University Hospital
Locations (1):
- Clinical Trial Center for Functional Foods Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided